CLINICAL TRIAL: NCT03682835
Title: The Effect of a Combination of Peppermint Oil and Caraway Oil on Gastric Motility, Nutrient Volume Tolerance, Gastric Emptying and Gastrointestinal Hormones in Healthy Volunteers
Brief Title: Effect of POCO on Gastric Function in HV
Acronym: POCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: POCO-study
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: gastric motility; gastric emptying; nutrient volume tolerance; peppermint oil; caraway oil

STUDY DESIGN:
Intervention Model Description: randomized, parallel, single-blind, placebo-controlled
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo treatment arm (Placebo Comparator): Placebo: 2 capsules per dose, 2 doses per study day.
  Interventions: Other: Placebo
- POCO treatment arm (Experimental): FDGard Capsule containing a combination of peppermint oil (41,5mg) and caraway oil (50mg); 2 capsules per dose, 2 doses per study day.
  Interventions: Dietary Supplement: FDGard

INTERVENTIONS:
Dietary Supplement: FDGard — capsule containing peppermint oil and caraway oil
  Arms: POCO treatment arm
Other: Placebo — Placebo capsule containing cellulose
  Arms: Placebo treatment arm

SUMMARY:
This study aims to investigate changes in gastric motility (including gastric accommodation), nutrient volume tolerance, gastric emptying and gastrointestinal hormones in healthy volunteers after an acute intake of a combination of peppermint oil and caraway oil, compared to placebo. In addition, the effect of a combination of peppermint oil and caraway oil on appetite-related sensations and upper gastrointestinal symptoms will be assessed.

Gastric emptying rate will be assessed using a 13C breath test. Intragastric pressure (IGP) will be measured using high-resolution manometry in fasted state and during intragastric infusion of a nutrient drink (350 mL or until full satiation). Appetite-related sensations and gastrointestinal symptoms were rated during IGP measurements. Blood samples were collected to assess peptide hormone levels.

DETAILED DESCRIPTION:
This study aims to investigate changes in gastric motility (including gastric accommodation), nutrient volume tolerance, gastric emptying and gastrointestinal hormones in healthy volunteers after an acute intake of a combination of peppermint oil and caraway oil, compared to placebo. In addition, the effect of a combination of peppermint oil and caraway oil on appetite-related sensations and upper gastrointestinal symptoms will be assessed. These outcomes will be studied on 2 study days. On study day 1, gastric emptying rate will be assessed using a 13C breath test 30 minutes after intake of study medication. This test is followed by an intragastric pressure (IGP) measurement during which 350 mL of a nutrient drink will be intragastrically infused 30 minutes after intake of study medication. On the second study day, IGP will be measured in fasted state for 4 hours after intake of study medication. Hereafter, a second dose of study medication will be administered. Thirty minutes later, a nutrient drink will be infused until the participant is fully satiated. Appetite-related sensations and gastrointestinal symptoms will be rated during IGP measurements on a 100mm VAS. Blood samples will be collected to assess peptide hormone levels.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female between 18 and 50 of age.
* Subject has a BMI between 20 and 25 and has a stable body weight for at least 3 consecutive months at start of study and no history of behavioral, therapeutic or surgical treatment aiming at or leading to weight loss/gain.
* Women of child-bearing potential agree to apply during the entire duration of the trial a highly effective method of birth control, which is defined as those which result in a low failure rate (i.e., less than 1% per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method, or some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 year without spontaneous menses.
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.

Exclusion Criteria:

* Subject is under age of legal consent, pregnant or breastfeeding.
* Subject with a BMI ≤ 20 or BMI ≥ 25.
* Subject has current symptoms or a history of gastrointestinal or other significant somatic or psychiatric diseases or drug allergies.
* Subject has a significant heart, lung, liver or kidney disease.
* Subject has any history of a neurological disorder.
* Subject has a history of abdominal surgery. Those having undergone a simple appendectomy more than 1 year prior to the screening visit may participate.
* History or current use of drugs that can affect gastrointestinal function, motility or sensitivity or gastric acidity.
* History or current use of centrally acting medication, including antidepressants, antipsychotics and/or benzodiazepines (in the last year before screening visit).
* Subject consumes excessive amounts of alcohol, defined as >14 units per week for women and >21 units per week for men.
* Subject is currently (defined as within approximately 1 year of the screening visit) a regular or irregular user (including "recreational use") of any illicit drugs (including marijuana) or has a history of drug (including alcohol) abuse. Further, patient is unwilling to refrain from the use of drugs during this study.
* High caffeine intake (> 500 ml coffee daily or equivalent).
* Inability or unwillingness to perform all of the study procedures, or the subject is considered unsuitable in any way by the principal investigator.
* Recent participation (<30 days) or simultaneous participation in another clinical study.
* Radiation exposure exceeding 1mSv during the last year (from other studies or medical procedures).
* Subject has had a PET-scan or CT-scan in the last year.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Gastric motility | Fed state: until 2 hours after the start of the liquid meal. Liquid meal started 30 minutes after POCO/placebo intake. Fasted state: until 4h after intake of POCO/placebo.
  motility of the stomach, including gastric accommodation

SECONDARY OUTCOMES:
Gastric emptying | Breath samples were collected before intake of medication/placebo and every 15 minutes until 4h after intake of 13C-octanoid acid
  Gastric emptying was assess by a 13C-octanoid acid breath test
Gastrointestinal symptoms | assessment by questionnaire (100 mm Visual Analogue Scale) every 15 minutes, until the end of the intragastric pressure measurement
  Change in subjective gastrointestinal symptom scores measured by visual analogue scale of 100 mm
Gastrointestinal peptide hormone levels | Hormone levels were assessed before and every 15 minutes after intake of POCO/placebo until the end of the intragastric pressure measurement
  change in gastrointestinale hormone levels induced by POCO intake

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, Principal Investigator — UZ Leuven / KU Leuven
Locations (1):
- TARGID, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No